CLINICAL TRIAL: NCT06746883
Title: A Single-arm, Open-label, Prospective, Observational Study to Assess the Safety of Sulbactam-durlobactam, Including the Risk of Hypersensitivity Reactions (Including Anaphylaxis) in Participants With Acinetobacter Baumannii-calcoaceticus Complex Infection
Brief Title: A Study to Assess the Safety and Risk of Hypersensitivity Reactions of Sulbactam-durlobactam in Adults With Acinetobacter Baumannii-calcoaceticus (ABC) Complex Infection
Status: Recruiting | Type: Observational
Sponsor: Innoviva Specialty Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CS2514-2023-003
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acinetobacter Baumannii-calcoaceticus Complex Infection (ABC)
Keywords: ABC infection; Acinetobacter baumannii-calcoaceticus complex infection; Hospital-acquired bacterial pneumonia; Ventilator-associated bacterial pneumonia; Sulbactam-durlobactam; Acinetobacter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Acinetobacter baumannii-calcoaceticus complex (ABC): Hospitalized participants with a proven or strongly suspected ABC infection who have received sulbactam-durlobactam as standard of care.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
The goal of this observational study is to evaluate the safety of sulbactam-durlobactam, as well as the risk of hypersensitivity reactions (including anaphylaxis) in participants with Acinetobacter baumannii-calcoaceticus complex infection. Participants will be followed for approximately 28 days in order to collect safety and reaction data.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥18 years old at the time of written informed consent and is hospitalized.
* Participant has provided the written informed consent. If a participant is unable to provide written informed consent due to their medical condition, the participant's legally authorized representative may consent on behalf of the participant, or the decision can be made according to the procedure permitted by local law and institutional standard operating procedures (SOPs).
* Participant has a proven or strongly suspected diagnosis of an infection caused by susceptible ABC isolates, based on investigator's clinical judgment.
* Participant initiates treatment with SUL-DUR per routine clinical care. Participants who receive SUL-DUR within 24 hours prior to enrollment are also eligible to participate. The decision to treat the participant with SUL-DUR is made prior to and independently of study participation.
* The participant has an expected survival of >48 hours at the time of written informed consent.

Exclusion Criteria:

* A history of significant hypersensitivity or allergic reaction to any β-lactam, or any contraindication to the use of β-lactam antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized participants
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing Treatment Emergent Adverse Events (TEAEs) defined as any event after exposure to sulbactam-durlobactam (SUL-DUR), or event already present that worsens in either intensity or frequency after exposure | 28 days
Number of participants experiencing TEAEs | 28 days
Incidence of maximum severity level of TEAEs | 28 days
Incidence of related TEAEs as assessed by the investigator. | 28 days
Incidence of serious TEAEs | 28 days
Percentage of participants experiencing Adverse Events of Special Interest (AESIs) defined as an AE or SAE of concern specific to the sponsor, for which ongoing monitoring is needed. AESIs include: Hypersensitivity reactions, including anaphylaxis. | 28 days
Number of participants experiencing AESIs | 28 days
Incidence of maximum severity level of AESIs | 28 days
Incidence of related AESIs as assessed by the investigator | 28 days
Incidence of serious AESIs | 28 days

SECONDARY OUTCOMES:
Actual observed values over time of liver function tests | Baseline and Day 28
Change from baseline values of liver function tests | Day 28
Actual observed values over time of systolic blood pressure | Baseline and Day 28
Change from baseline values over time of systolic blood pressure | Day 28
Actual observed values over time of diastolic blood pressure | Baseline and Day 28
Change from baseline values of diastolic blood pressure | Day 28
Actual observed values over time of temperature | Baseline and Day 28
Change from baseline values of temperature | Day 28
Actual observed values over time of pulse rate | Baseline and Day 28
Change from baseline values of pulse rate | Day 28
Actual observed values over time of respiration rate | Baseline and Day 28
Change from baseline values of respiration rate | Day 28
Summary of observed values over time of ECG QT measurements | Baseline and Day 28
Change from baseline values over time of ECG QT measurements | Day 28
Summary of observed values over time of hemoglobin | Baseline and Day 28
Change from baseline values over time of hemoglobin | Day 28
Summary of observed values over time of white blood count | Baseline and Day 28
Change from baseline values over time of white blood count | Day 28
Summary of observed values over time of platelets | Baseline and Day 28
Change from baseline values over time of platelets | Day 28

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Kansas Medical Center-Kansas City-3901 Rainbow Blvd, Kansas City, Kansas
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Ochsner LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Montefiore Medical Group Family Care Center, The Bronx, New York
  - Summa Health System - Akron - 75 Arch Street, Akron, Ohio
  - The Carl and Edyth Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Prisma Health - Infectious Diseases - Greenville, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified IPD may be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests may be submitted starting 6 months after primary article publication and the data will be made accessible for up to 24 months; extensions may be considered on a case-by-case basis.
Access Criteria: Subject to certain criteria, conditions, and exceptions and upon completion of the review and approval of the Research Proposal and Statistical Analysis Plan, Qualified Researchers engaging in independent scientific research can be provided de-identified IPD following the execution of a Data Sharing Agreement.
URL: http://clinicaltrials@ISTX.com